CLINICAL TRIAL: NCT06089096
Title: Exploring the Association of Sleep Apnea With Cognitive Function in Subjects With Subjective or Mild Cognitive Impairment
Brief Title: Sleep Apnea and Cognitive Function in Subjects With Subjective or Mild Cognitive Impairment
Status: Recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Mary Ip Sau-man, Honorary Clinical Professor, The University of Hong Kong
Other Study IDs: UW 23-072
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Obstructive Sleep Apnea; Mild Cognitive Impairment; Subjective Cognitive Impairment
MeSH Terms: conditions — Sleep Apnea, Obstructive; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MCI or SCI patient: At baseline: Cognitive tests, questionnaire, and Home Sleep Apnea Test will be done.
  Interventions: Diagnostic Test: Home Sleep Apnea test (HSAT)

INTERVENTIONS:
Diagnostic Test: Home Sleep Apnea test (HSAT) — Patient will received HSAT at baseline

SUMMARY:
Obstructive sleep apnea (OSA) is recurrent episodes of partial or complete obstruction of the upper airway during sleep that causes intermittent hypoxia and sleep fragmentation and leads to cardiometabolic and neurocognitive sequelae. Chronic intermittent hypoxia, sleep fragmentation of OSA, and insufficient sleep have been significantly associated with higher risks of neurocognitive impairment, including mild cognitive impairment (MCI) and Alzheimer's disease. Thus, sleep and circadian function might be modifiable neurocognitive impairment factors.

The significance of the study is to understand the relationships of MCI with sleep apnea and sleep-related symptoms, which helps pave the groundwork for further research.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is recurrent episodes of partial or complete obstruction of the upper airway during sleep that causes intermittent hypoxia and sleep fragmentation. Chronic intermittent hypoxia, sleep fragmentation of OSA, and insufficient sleep have been significantly associated with higher risks of neurocognitive impairment, including mild cognitive impairment (MCI) and Alzheimer's disease. Thus, sleep and circadian function might be modifiable neurocognitive impairment factors.

A recent review of 11 studies involving 5826 subjects [96% with OSA and 9% with MCI or Alzheimer's disease] suggests OSA is a modifiable risk factor for cognitive decline. Thus, improving sleep, sleep apnea and circadian function could be a high-value intervention target to alleviate cognitive impairment and decline in subjects with MCI.

The study aims to understand the relationships of prevalent sleep apnea and sleep-related symptoms with neurocognitive status in patients who presented with the main complaint of neurocognitive impairment ( to the Memory clinic). The information would help pave the groundwork for further research.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above
* Clinical diagnosis of mild cognitive impairment (MCI) based on Petersen's criteria. The criteria include the following: (1) memory problems, (2) objective memory disorder, (3) absence of other cognitive disorders or repercussions on daily life, (4) normal general cognitive function and (5) absence of dementia OR,
* Diagnosis of subjective cognitive impairment, based on the subject's own complaint of cognitive impairment but with an unremarkable assessment of the Hong Kong version of Montreal Cognitive Assessment scores
* Able to speak and read Chinese
* Adequate visual and auditory to perform a cognitive test

Exclusion Criteria:

* Diagnosed psychiatric illness with or without medication, e.g. major depressive disorder.
* Other clear organic causes of cognitive impairment, e.g. old stroke, brain tumour, dementia with Lewy body, Parkinson's disease, normal pressure hydrocephalus, neurosyphilis, autoimmune encephalitis, substance abuse, history of alcohol abuse.
* Diagnosis of major unstable illness or cancer on active treatment
* Unable to perform Home Sleep Apnea Test
* Those patients who require legal guardians

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This cross-sectional study aims to recruit subjects with mild or subjective cognitive impairment in Queen Mary Hospital, Hong Kong.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Sleep study parameters | Baseline
  Measured by Apnea Hypopnea Index (AHI). Score less than 5 is no OSA, score 5-15 is categorized as mild OSA, 15-30 is categorized as moderate OSA, and>30 is severe OSA.

SECONDARY OUTCOMES:
Daytime sleepiness | Baseline
  Measured by Epworth Sleepiness Scale. Each item asks the individual to rate their daytime sleepiness. The total score ranges from 0 to 24. The higher the scores, the greater the severity of daytime sleepiness
Sleep apnea symptoms | Baseline
  Measured by Pittsburgh Sleep Quality Index. Each of the sleep components yields a score ranging from 0 to 3, with 3 indicating the greatest dysfunction. The sleep component scores are summed to yield a total score ranging from 0 to 21, with the higher total score indicating worse sleep quality.
Insomnia symptoms | Baseline
  Measured by Severe Insomnia Index. Each item asks the individual to rate the severity of his or her symptoms with a 4-point Likert scale. The total score ranges from 0 to 28. The higher the scores the greater the severity of insomnia
Sleep profile and quality | Baseline
  Measured by Pittsburgh Sleep Quality Index. Each of the sleep components yields a score ranging from 0 to 3, with 3 indicating the greatest dysfunction. The sleep component scores are summed to yield a total score ranging from 0 to 21, with the higher total score indicating worse sleep quality.
Depression symptoms | Baseline
  Measured by Geriatric Depression Scale - short form. The score ranges from 0 to 15. The higher the scores the more severe of depression.
Activities of Daily Living | Baseline
  Measured by Instrumental Activities of Daily Living Scale (I.A.D.L.) and Simplified Barthel ADL index.
  The total score of I.A.D.L ranges from 0 to 8, "0" is the worst possible score, while "8" is the best possible score.
  The total score of A.D.L ranges from 0 to 20, "0" is the worst possible score, while "20" is the best possible score.
Cognitive function | Baseline
  Measured by Montreal Cognitive Assessment (MoCA) score and ADAS-Cog. The scores of MoCA range from 0 to 30, "0" is the worst possible score and "30" is the best possible score. The scores of ADAS-Cog range from 0 to 70, "0" is the best possible score and "70" is the worst possible score.
Ability to inhibit cognitive interference | Baseline
  Measured by Stroop Colour and Word Test (SCWT). Scored by time and error. A longer time indicates a worst score, while a shorter time indicates a better score.

CONTACTS AND LOCATIONS:
Overall Officials: Sau Man Mary Ip, MD, Principal Investigator — School of Clinical Medicine, The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yaffe K, Laffan AM, Harrison SL, Redline S, Spira AP, Ensrud KE, Ancoli-Israel S, Stone KL. Sleep-disordered breathing, hypoxia, and risk of mild cognitive impairment and dementia in older women. JAMA. 2011 Aug 10;306(6):613-9. doi: 10.1001/jama.2011.1115. PMID 21828324
- [Background] Emamian F, Khazaie H, Tahmasian M, Leschziner GD, Morrell MJ, Hsiung GY, Rosenzweig I, Sepehry AA. The Association Between Obstructive Sleep Apnea and Alzheimer's Disease: A Meta-Analysis Perspective. Front Aging Neurosci. 2016 Apr 12;8:78. doi: 10.3389/fnagi.2016.00078. eCollection 2016. PMID 27148046
- [Background] Leng Y, McEvoy CT, Allen IE, Yaffe K. Association of Sleep-Disordered Breathing With Cognitive Function and Risk of Cognitive Impairment: A Systematic Review and Meta-analysis. JAMA Neurol. 2017 Oct 1;74(10):1237-1245. doi: 10.1001/jamaneurol.2017.2180. PMID 28846764
- [Background] Musiek ES, Ju YS. Targeting Sleep and Circadian Function in the Prevention of Alzheimer Disease. JAMA Neurol. 2022 Sep 1;79(9):835-836. doi: 10.1001/jamaneurol.2022.1732. No abstract available. PMID 35816332